CLINICAL TRIAL: NCT06811597
Title: The Effects of Fixed Space Maintainers Luting with Self-Adhesive Resin Cement on the Gingival Crevicular Fluid of Interleukin-18 Level
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Özgür Doğan, Associate Professor, Afyonkarahisar Health Sciences University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2011-KAEK-2/ 2022/7336
Record Dates: First submitted 2025-01-24; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Gingival and Periodontal Disease; Space Maintenance; Resin Cements; Interleukin
Keywords: Fixed Space Maintainer; IL-18; Resin Cement; Self Adhesive; Gingival Inflammation; Luting Cement
MeSH Terms: conditions — Periodontal Diseases; Gingivitis

STUDY DESIGN:
Intervention Model Description: This split-mouth design study involved 31 children aged 6 to 10 years who prematurely lost their mandibular second primary molars. The left mandibular first molars were bonded with FSM High-Q-Bond Band™ self-adhesive resin cement, while the right molars were bonded with Meron (conventional glass ionomer cement). Gingival Index (GI), Plaque Index (PI), and Periodontal Probing Depth (PPD) were measured before luting and at the 1-week follow-up. Gingival crevicular fluid (GCF) was collected from the abutment teeth using Periopaper® strips before luting and at the one-week follow-up. ELISA was then performed to measure the levels of the proinflammatory cytokine Interleukin-18(IL-18).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Voco Meron Conventional Glass Ionomer Group (Active Comparator): The right molars were bonded with conventional glass ionomer cement.
  Interventions: Procedure: Voco Meron Conventional Glass Ionomer
- High-Q-Bond Band™ self-adhesive resin cement (Experimental): The left mandibular first molars were bonded with FSM High-Q-Bond Band™ self-adhesive resin cement.
  Interventions: Procedure: High-Q-Bond Band™ self-adhesive resin cement.

INTERVENTIONS:
Procedure: Voco Meron Conventional Glass Ionomer — The right molars were bonded with Meron
  Arms: Voco Meron Conventional Glass Ionomer Group
Procedure: High-Q-Bond Band™ self-adhesive resin cement. — The left mandibular first molars were bonded with FSM High-Q-Bond Band™ self-adhesive resin cement.
  Arms: High-Q-Bond Band™ self-adhesive resin cement

SUMMARY:
Background:In pediatric dentistry, fixed space maintainers are crucial for preserving the space in edentulous areas following premature tooth loss and promoting the healthy development of the dental arch, maxilla, and mandibula. A vital aspect in ensuring the long-term functionality of the space maintainer is the selection of the appropriate luting agent. Conventional glass ionomer cements (GIC), known for their chemical properties and biocompatibility, are widely regarded as safe and effective luting agents. Despite the prevalent use of resin cements (RCs) in modern dentistry, studies examining the effects of fixed space maintainers (FSMs) luted with resin cements (RCs) on periodontal status are lacking.

Material:This split-mouth design study involved 31 children aged 6 to 10 years who prematurely lost their mandibular second primary molars. The left mandibular first molars were bonded with FSM High-Q-Bond Band™ self-adhesive resin cement, while the right molars were bonded with Meron (conventional glass ionomer cement). Gingival Index (GI), Plaque Index (PI), and Periodontal Probing Depth (PPD) were measured before luting and at the 1-week follow-up. Gingival crevicular fluid (GCF) was collected from the abutment teeth using Periopaper® strips before luting and at the one-week follow-up. ELISA was then performed to measure the levels of the proinflammatory cytokine Interleukin-18(IL-18). Statistical Analyses involved the Mann-Whitney U test for comparing two groups of qualitative and quantitative variables, and the Wilcoxon Signed Ranks test for assessing differences between two dependent quantitative variables. A significance threshold of p < 0.05 was used for statistical inference.

DETAILED DESCRIPTION:
Introduction Fixed space maintainers (FSMs) are important preventive orthodontic devices used in pediatric dentistry. These devices are specifically designed to preserve the spaces left by premature tooth loss or planned tooth extractions. Maintaining these spaces is crucial for guiding the proper eruption of permanent teeth, contributing to a child's healthy dental development. Pediatric dentists are the most frequently consulted professionals during this stage, and their preventive practices significantly impact the preservation of the edentulous space during the transition from mixed dentition to permanent dentition.

The primary objective of all types of space maintainers in primary and mixed dentition is to preserve arch length by preventing space loss within the dental arch. Space loss may occur as a result of the mesial migration of teeth positioned distal to an edentulous area through tipping, or due to the distal drifting of teeth that remain mesial to the edentulous region. The type and design of space maintainers employed to preserve the edentulous spaces resulting from premature loss of primary teeth are contingent upon various factors. These factors include the number of teeth that have been lost in the affected area, the stage of the child's dental development, and the specific dental arch where the space maintainer is to be applied. Considering all these factors, FSMs are the most preferred option among the various types of space maintainers, as they remain unaffected by jaw or dental arch conditions.

Preventing malocclusions in a developing child due to the premature loss of primary teeth is crucial. This can be accomplished by using a space maintainer as soon as possible after a tooth extraction. This can protect the space left by the missing tooth and help maintain the proper arch length as the child continues to grow. FSMs need to remain cemented in the mouth for an extended period, as even a matter of days can be significant in this process. To achieve optimal results, the cementation process must be conducted with durable luting cement. Traditionally, it has been advised to cement FSMs using conventional glass ionomer cement (GIC). However, over the past decade, resin cement (RC) has become increasingly prevalent due to significant advancements in bonding technology and the rising adoption of adhesive resin cement within dentistry.

While resin cement has been employed to enhance the survival of FSMs, it is crucial to note that research investigating periodontal inflammation in children arising from residual cement following the FSM cementation process is lacking. Numerous inflammatory cytokine biomarkers indicate the presence of gingival inflammation. Pro-inflammatory cytokines, tumor necrosis factor(TNF-α), anti-inflammatory cytokines, and host factor metalloproteinases play significant roles in regulating inflammatory responses. Interleukin-18 (IL-18) is a significant pro-inflammatory cytokine belonging to the Interleukin-1 (IL-1) family. It is essential in the immune response to infections and various diseases. The function of IL-18 in the inflammatory response is to facilitate the expression of adhesion molecules on endothelial cells, thereby increasing the recruitment of immune cells to the site of inflammation. The accumulation of IL-18 in regions that are persistently exposed to irritants triggers chronic tissue damage, facilitating the progression of the disease's pathogenesis. The role of IL-18 in immune regulation and inflammation suggests that it may serve as a potential biomarker for tracking the progression of various diseases. Studies have indicated that the expression levels of IL-18 are significantly elevated in gingival crevicular fluid and gingival tissue samples associated with gingival inflammation and periodontal diseases.

Gingival crevicular fluid (GCF) is recognized as the primary medium for analyzing alterations in the local tissue environment, thereby facilitating the assessment of periodontal health and disease. This fluid is instrumental in understanding the physiological changes occurring in periodontal conditions. The noninvasive collection of biomarkers in GCF is an essential diagnostic method for accurately assessing gingival health in clinical settings.

Upon re-evaluating the FSM treatment protocol in light of this information, it becomes clear that FSMs are frequently cemented within the gingival pocket in cases where they come into contact with the gingiva. Current literature remains unclear about inflammation effects in the periodontal sulcus caused by the use of resin cement for luting space maintainers. The null hypothesis of this study posits that FSMs luted with conventional GIC and those luted with resin cement result in identical alterations in IL-18 levels within the GCF of pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children who have not received any antibiotic treatment in the past four months,
* Children who do not have any underlying systemic diseases.
* Children who are not required to take medication regularly,
* Both girls and boys between the ages of 6 and 10.
* The second primary molar teeth (75 and 85) were extracted from patients due to caries and associated periapical pathologies.
* The presence of the succeeding tooth germ.
* Pediatric patients exhibiting Angle Class I occlusal relationships.
* Children without skeletal abnormalities.
* Existence of the antagonistic tooth of the abutment tooth.
* Children and their parents willing to participate in the study and attend the control session one week later were included.

Exclusion Criteria:

* The patient presents with periodontal disease.
* Children with cognitive disabilities, including autism and attention deficit hyperactivity disorder, as well as those with mental health conditions such as cerebral palsy and Down syndrome.
* Children and their parents who did not meet the specified criteria were excluded from the study.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
IL-18 | 1 week.
  We will examine IL-18 expression levels and changes in gingival crevicular fluid and gingival tissue samples related to gingivitis and periodontal diseases.

SECONDARY OUTCOMES:
Plaque İndex | 1 week
  The plaque index measures the amount of plaque accumulated in the periodontium area where the assessment is made. The plaque buildup caused by the fixed space maintainer will be assessed.
Gingival Index | 1 week
  The gingival index is one of the evaluation criteria of periodontal health.
Periodontal Probing Depth | 1 week
  It indicates whether the gingivitis has spread to the alveolar bone. The cause of the inflammation caused by the fixed space maintainer will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Suat Serhan Altıntepe Doğan, Assoc. Prof. (PhD), Study Director — Afyonkarahisar Health Sciences University
Locations (2):
- Turkey (Türkiye) (2):
  - Afyonkarahisar Health Sciences University, Afyonkarahisar
  - Afyonkarahisar Health Science, Afyonkarahisar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cengiz A, Karayilmaz H. Comparative evaluation of the clinical success of 3D-printed space maintainers and band-loop space maintainers. Int J Paediatr Dent. 2024 Sep;34(5):584-592. doi: 10.1111/ipd.13159. Epub 2024 Jan 12. PMID 38217333
- [Background] Dinarello CA. Interleukin 1 and interleukin 18 as mediators of inflammation and the aging process. Am J Clin Nutr. 2006 Feb;83(2):447S-455S. doi: 10.1093/ajcn/83.2.447S. PMID 16470011
- [Background] Johnson RB, Serio FG. Interleukin-18 concentrations and the pathogenesis of periodontal disease. J Periodontol. 2005 May;76(5):785-90. doi: 10.1902/jop.2005.76.5.785. PMID 15898940
- [Background] Jablonska E, Izycka A, Jablonska J, Wawrusiewicz N, Piecuch J. Role of IL-18 in the secretion of Il-1beta, sIL-1RII, and IL-1Ra by human neutrophils. Immunol Invest. 2001 Aug;30(3):221-9. doi: 10.1081/imm-100105066. PMID 11570642
- [Background] Orozco A, Gemmell E, Bickel M, Seymour GJ. Interleukin-1beta, interleukin-12 and interleukin-18 levels in gingival fluid and serum of patients with gingivitis and periodontitis. Oral Microbiol Immunol. 2006 Aug;21(4):256-60. doi: 10.1111/j.1399-302X.2006.00292.x. PMID 16842511
- [Background] Nair V, Grover V, Arora S, Das G, Ahmad I, Ohri A, Sainudeen S, Saluja P, Saha A. Comparative Evaluation of Gingival Crevicular Fluid Interleukin-17, 18 and 21 in Different Stages of Periodontal Health and Disease. Medicina (Kaunas). 2022 Aug 3;58(8):1042. doi: 10.3390/medicina58081042. PMID 36013509
- [Background] Kinney JS, Morelli T, Oh M, Braun TM, Ramseier CA, Sugai JV, Giannobile WV. Crevicular fluid biomarkers and periodontal disease progression. J Clin Periodontol. 2014 Feb;41(2):113-120. doi: 10.1111/jcpe.12194. Epub 2013 Dec 12. PMID 24303954
- [Background] Kaur J, Singh A, Sadana G, Mehra M, Mahajan M. Evaluation of Shear Peel Bond Strength of Different Adhesive Cements Used for Fixed Space Maintainer Cementation: An In Vitro Study. Int J Clin Pediatr Dent. 2021 Mar-Apr;14(2):175-179. doi: 10.5005/jp-journals-10005-1932. PMID 34413586
- [Background] Ierardo G, Luzzi V, Lesti M, Vozza I, Brugnoletti O, Polimeni A, Bossu M. Peek polymer in orthodontics: A pilot study on children. J Clin Exp Dent. 2017 Oct 1;9(10):e1271-e1275. doi: 10.4317/jced.54010. eCollection 2017 Oct. PMID 29167720
- [Background] Khanna S, Rao D, Panwar S, Pawar BA, Ameen S. 3D Printed Band and Loop Space Maintainer: A Digital Game Changer in Preventive Orthodontics. J Clin Pediatr Dent. 2021 Jul 1;45(3):147-151. doi: 10.17796/1053-4625-45.3.1. PMID 34192758
- [Background] Neto HNM, Leite JVC, de Medeiros JM, E Silva Campos D, de Araujo Ferreira Muniz I, De Andrade AKM, Duarte RM, De Souza GM, Lima RBW. Scoping review: Effect of surface treatments on bond strength of resin composite repair. J Dent. 2024 Jan;140:104737. doi: 10.1016/j.jdent.2023.104737. Epub 2023 Oct 8. PMID 37816488
- [Background] Anumula L, Ramesh S, Kolaparthi VSK. Matrix metalloproteinases in dentin: Assessing their presence, activity, and inhibitors - a review of current trends. Dent Mater. 2024 Nov;40(11):2051-2073. doi: 10.1016/j.dental.2024.09.011. Epub 2024 Oct 5. PMID 39368893
- [Background] Barathi D, Jampanapalli SR, Patloth T, Konda S, Inguva H, Shaik H. Comparative Evaluation of Shear Bond Strength of Bonded Space Maintainers Using Ormocers, Nanofilled and Glass Fiber-reinforced Adhesive Composites. Int J Clin Pediatr Dent. 2024 Jun;17(6):695-701. doi: 10.5005/jp-journals-10005-2904. PMID 39391145
- [Background] Alvarenga M, Machado L, Prado A, Veloso S, Monteiro G. Self-adhesive resin cement versus conventional cements on the failure rate of indirect single-tooth restorations: A systematic review and meta-analysis of randomized clinical trials. J Prosthet Dent. 2024 Nov;132(5):880.e1-880.e8. doi: 10.1016/j.prosdent.2024.04.027. Epub 2024 May 25. PMID 38797576
- [Background] Hemdan ME, El Kalla IHH, El Agamy RA. Clinical Evaluation of Different Designs of Fixed Space Maintainer: A Randomized Clinical Trial. Int J Clin Pediatr Dent. 2024 Apr;17(4):442-450. doi: 10.5005/jp-journals-10005-2835. PMID 39144172
- [Background] Laing E, Ashley P, Naini FB, Gill DS. Space maintenance. Int J Paediatr Dent. 2009 May;19(3):155-62. doi: 10.1111/j.1365-263X.2008.00951.x. PMID 19385999
- [Background] Gupta A, Dutta B, Dhull KS, Md I, Wandile B. A Leap Beyond Traditional Methods: A Case Report on the Horizontal Loop Distal Shoe. Cureus. 2024 May 6;16(5):e59724. doi: 10.7759/cureus.59724. eCollection 2024 May. PMID 38840994
- [Background] Qudeimat MA, Sasa IS. Clinical success and longevity of band and loop compared to crown and loop space maintainers. Eur Arch Paediatr Dent. 2015 Oct;16(5):391-6. doi: 10.1007/s40368-015-0183-y. Epub 2015 Mar 19. PMID 25788173
- [Background] Qudeimat MA, Fayle SA. The longevity of space maintainers: a retrospective study. Pediatr Dent. 1998 Jul-Aug;20(4):267-72. PMID 9783298
- [Background] Lee JH. Fully digital workflow for the fabrication of a tooth-colored space maintainer for a young patient. J Esthet Restor Dent. 2023 Jun;35(4):561-566. doi: 10.1111/jerd.12939. Epub 2022 Jun 22. PMID 35731166
- [Background] Barros SE, Siqueira SP, Janson G, Chiqueto K. Short-term efficacy of vacuum-formed maintainer for deciduous second molar space maintenance in the mixed dentition: A single-centre, randomized controlled clinical trial. Orthod Craniofac Res. 2021 Nov;24(4):502-510. doi: 10.1111/ocr.12460. Epub 2021 Jan 4. PMID 33352006
- [Background] Heidari A, Mokhtari S, Hamrah MH, Tavana Z, Heydarigoojani M, Tavana N. Investigating the Factors Affecting the Need for Unilateral Space Maintainer for First Primary Molars in Late Mixed Dentition. Biomed Res Int. 2022 Mar 29;2022:7604144. doi: 10.1155/2022/7604144. eCollection 2022. PMID 35392262
- [Background] Dogan O, Dogan SSA. Arm design of band and loop space maintainer affects its longevity: a patient-specific finite element study. J Clin Pediatr Dent. 2024 Jan;48(1):171-183. doi: 10.22514/jocpd.2024.019. Epub 2024 Jan 3. PMID 38239170
- [Background] Watt E, Ahmad A, Adamji R, Katsimpali A, Ashley P, Noar J. Space maintainers in the primary and mixed dentition - a clinical guide. Br Dent J. 2018 Aug 24;225(4):293-298. doi: 10.1038/sj.bdj.2018.650. PMID 30141512
- [Background] Nascimento EB, Rodrigues R, Manso MC. Prevalence of dental floss use in deciduous dentition: A systematic review and meta-analysis. Int J Dent Hyg. 2023 Feb;21(1):116-127. doi: 10.1111/idh.12611. Epub 2022 Aug 15. PMID 35924390
- [Background] Law CS. Management of premature primary tooth loss in the child patient. J Calif Dent Assoc. 2013 Aug;41(8):612-8. PMID 24073500